CLINICAL TRIAL: NCT06738394
Title: Enhancing Physical Function in Older Adults With Chronic Kidney Disease (EPIC): A Pilot Randomized Controlled Trial
Brief Title: Enhancing Physical Function in Older Adults With Chronic Kidney Disease
Acronym: EPIC
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Wake Forest University Health Sciences (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IRB00118658
Record Dates: First submitted 2024-12-12; First posted 2024-12-17 (Actual); Last update posted 2025-12-31 (Actual); Status verified 2025-09

CONDITIONS: Chronic Kidney Diseases
Keywords: kidney disease; resistance training; older adults
MeSH Terms: conditions — Renal Insufficiency, Chronic; Kidney Diseases | interventions — Neuropsychological Tests

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High-Velocity Resistance Training (HVRT) (Experimental): Those assigned to HVRT will attend three small-group (two to five people) exercise sessions lasting 60-75 minutes per week consisting of upper- and lower-body movements performed with weighted vests, medicine balls, and resistance bands. For all exercises, the concentric phase (muscle-shortening portion) will be performed as quickly as possible while maintaining good form, followed by a 1-second pause and then the eccentric phase (lengthening portion) completed in a slow and controlled fashion. Following completion of the 12-week intervention, all participants will be asked to complete the same baseline tests to assess changes in physical function, body composition, quality of life, and cognitive function outcomes.
  Interventions: Behavioral: High-Velocity Resistance Training
- Control Group (Active Comparator): Participants randomized to the attention control group will receive dedicated contact, information, and motivation throughout the course of the intervention via weekly group sessions and informational handouts. Each in-person group meeting will last approximately one hour. These group sessions will take place in a classroom/conference room setting and include information on such topics as blood pressure, reading food labels, healthy eating, and memory. The class will be a PowerPoint presentation with incorporated question/answer, lively discussion, and group-bonding activities. Following completion of the 12-week intervention, all participants will be asked to complete the same baseline tests to assess changes in physical function, body composition, quality of life, and cognitive function outcomes.
  Interventions: Behavioral: Attention

INTERVENTIONS:
Behavioral: High-Velocity Resistance Training — High-velocity resistance training for patients with non-dialysis dependent chronic kidney disease Stages 3-5 with mobility limitations.
  Arms: High-Velocity Resistance Training (HVRT)
Behavioral: Attention — Dedicated contact, information, and motivation throughout the course of the study via weekly group sessions and informational handouts.
  Arms: Control Group

SUMMARY:
The goal of this pilot randomized controlled trial is to examine the feasibility and safety of a 12-week high-velocity resistance training (HVRT) intervention in older adults with chronic kidney disease (CKD) stages 4-5 and to generate preliminary data to inform a future study investigating the efficacy of HVRT for improving muscle power and physical function. Researchers will compare HVRT to an attention control condition consisting of weekly group sessions covering topics on healthy lifestyle. This study seeks to:

1. Determine whether implementing an HVRT intervention is feasible and safe for mobility-limited older adults with advanced CKD.
2. Collect preliminary data on the efficacy of HVRT for improving muscle power and physical function in mobility-limited older adults with advanced CKD.

DETAILED DESCRIPTION:
Older adults with advanced chronic kidney disease (CKD) commonly exhibit severe impairments in physical function (i.e., inability to perform activities of daily living). Muscle power-the product of muscle force and velocity of contraction- is now widely considered to be a critical determinant of physical function in older adults. Despite this, muscle power has been largely overlooked in the aims and outcomes of exercise interventions for patients with CKD. Several clinical trials have shown that high-velocity resistance training (HVRT) programs consisting of functional movements performed "as fast as possible" with low external loads are safe and effective for improving muscle power and physical function in older adults. However, the available evidence on the effects of exercise interventions designed to improve muscle power in patients with CKD is scarce. This study seeks to determine whether an HVRT intervention in mobility-limited older adults with advanced CKD is feasible, safe, and potentially effective for improving muscle power and physical function.

ELIGIBILITY:
Inclusion Criteria:

* Chronic kidney disease stages 3-5
* Capacity to complete physical exercise
* Lives within 20 miles of Wake Forest Reynolda Campus
* Fluent English speaker
* Does not plan to travel outside of home area for an extended period of time during study
* Willing to be randomized to either intervention group

Exclusion Criteria:

* Receiving renal replacement therapy (e.g. hemodialysis, peritoneal dialysis) or anticipated to start renal replacement therapy in the next 6 months
* Dependent on a wheelchair
* Current participation in a resistance training program
* Joint replacement or orthopedic surgery in the previous 6 months or planning to have surgery in the next 6 months months
* Absolute contraindications to exercise testing according to ACSM:

Acute myocardial infarction within the past 6 months Ongoing unstable angina Uncontrolled cardiac arrhythmia with hemodynamic compromise Active endocarditis Symptomatic severe aortic stenosis Decompensated heart failure Acute pulmonary embolism, pulmonary infarction, or deep venous thrombosis Acute myocarditis or pericarditis Acute aortic dissection

* Parkinson's disease
* Respiratory disease requiring oxygen
* Cancer requiring treatment
* Currently receiving physical therapy or cardiopulmonary rehabilitation
* Type I or insulin dependent Type II Diabetes
* Scoring below 32 points on the Telephone Interview for Cognitive Status (TICS)
* Site PI/Study Clinician discretion regarding medical status, appropriateness of participation or concern about intervention adherence

Ages: 65 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-07-31 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Number of Participants Enrolled | Month 6
  Number of participants enrolled with a goal of 30.
Percent of Participant Adherence | Week 13
  Percentage of exercise sessions attended for the HVRT group (out of 36 total exercise sessions)
Percent of Participant Retention | Week 13
  Percentage of participants retained at the final follow visit.

SECONDARY OUTCOMES:
Change in Short Physical Performance Battery (SPPB) Score | From baseline to Follow-up (Week 13)
  The short physical performance battery (SPPB) consists of three tests to assess lower extremity function: a balance test, a gait speed test, and a sit-to-stand test. Performance in each test will be assigned a score ranging from 0 to 4 points, and these scores will be summed to calculate the SPPB score out of 12. A higher SPPB score indicates better function, and scores of 10 or lower are indicative of high risk of disability.
Change in Timed Up and Go Test duration | From baseline to Follow-up (Week 13)
  For the timed up-and-go test, the time to complete this task will be measured in seconds. A lower number of seconds to complete the task is indicative of higher physical function.
Change in lower body peak power | From baseline to Follow-up (Week 13)
  Leg press peak power will be assessed at 5 relative intensities (40%, 50%, 60%, 70%, and 80% 1-repetition maximum). The highest peak power measurement among those 5 loads will be recorded as peak power. Greater peak power is indicative of greater lower body neuromuscular function.

OTHER OUTCOMES:
Change in Appendicular Lean Mass | From baseline to Follow-up (Week 13)
  Appendicular Lean Mass (kg/m^2) will be measured via dual-energy X-ray absorptiometry (DXA). Higher appendicular lean mass is indicative of improved body composition.
Change in isometric leg extension strength | From baseline to Follow-up (Week 13)
  Isometric leg extension strength will be measured with a maximal isometric voluntary contraction of the dominant leg knee extensor muscles using a MicroFET2 hand-held dynamometer. Greater peak force is indicative of greater knee extensor strength.
Change in lower body strength | From baseline to Follow-up (Week 13)
  Lower body strength will be measured as the 1-repetition maximum on the leg press, which is the maximum load (kg) that can be moved 1 time only throughout the full range of motion. Increase in leg press 1-repetition maximum is indicative of improved lower body strength.
Change in lower body muscle endurance | From baseline to Follow-up (Week 13)
  Lower body muscle endurance will be measured on the leg press as the maximum number of repetitions completed at a load of 70% of baseline 1-repetition maximum with a fixed cadence of 60 bpm. An increase in the number of repetitions completed is indicative of an improvement in lower body muscle endurance.
Change in muscle activation | From baseline to Follow-up (Week 13)
  Muscle activation of knee extensors (rectus femoris, vastus medialis, and vastus lateralis) will be assessed by surface electromyography (EMG) during the maximal voluntary contraction (MVC) and during the leg press exercise testing. An increase in the peak EMG root-mean-square amplitude relative to the amplitude during MVC (%MVC) is indicative of greater muscle activation.
Change in average daily steps | From baseline to Follow-up (Week 13)
  An ActivPAL 4 triaxial accelerometer will be worn on the midline of the non-dominant thigh for 7 consecutive days prior to the start of the intervention and during the final week of the intervention. An increase in the average number of steps per day is indicative of increased physical activity level.
Change in average daily minutes spent sedentary | From baseline to Follow-up (Week 13)
  The average number of minutes spent in sedentary behavior per day will be measured with an ActivPAL 4 triaxial accelerometer. An decrease in the average number of minutes spent in sedentary behavior per day is indicative of a decrease in sedentary activity.
Change in average daily minutes spent stepping | From baseline to Follow-up (Week 13)
  The average number of minutes spent stepping per day will be measured with an ActivPAL 4 triaxial accelerometer. An increase in the number of minutes spent stepping per day is indicative of an increase in physical activity.
Change in average daily minutes spent stepping above 75 steps per minute and 100 steps per minute | From baseline to Follow-up (Week 13)
  The average number of minutes spent stepping above 75 steps per minute and 100 steps per minute per day will be measured with an ActivPAL 4 triaxial accelerometer. An increase in the number of minutes spent stepping above 75 steps per minute and 100 steps per minute is indicative of an increase in moderate-to-vigorous intensity physical activity.
Change in Symbol Digit Coding Test Score | From baseline to Follow-up (Week 13)
  The Symbol Digit Coding Test measures complex information processing accuracy, complex attention, visual-perceptual speed, and information processing speed. The score is the number of correct symbols drawn within a period of 120 seconds. One point is given for each correctly drawn symbol completed within the time limit. The maximum score is 133.
  High scores indicate higher cognitive functioning.
Change in Four-Part Continuous Performance | From baseline to Follow-up (Week 13)
  The 4PCPT test is a four-part test that measures a subject's working memory and sustained attention. Higher scores indicate higher cognitive functioning.
Change in Shifting Attention Test Score | From baseline to Follow-up (Week 13)
  SAT test is a measure of ability to shift from one instruction set to another quickly and accurately. Higher scores indicate higher cognitive functioning.
Change in Stroop Test Score | From baseline to Follow-up (Week 13)
  Stroop test has three parts. Higher scores indicate higher cognitive functioning.
Change in Kidney Disease Quality of Life Short Form (KDQOL-SF) Scores | From baseline to Follow-up (Week 13)
  The KDQOL-SF version 1.3 is a self-report measure developed for individuals with kidney disease. It includes 43 kidney-disease targeted items as well as 36 items that provide a generic core and an overall health rating item. 0-100 possible range, with higher scores always reflecting better quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Eliott Arroyo, PhD, Principal Investigator — Wake Forest University Health Sciences
Locations (1):
- Wake Forest University Health Sciences, Winston-Salem, North Carolina, United States

IPD SHARING:
Plan to Share IPD: No